CLINICAL TRIAL: NCT03958669
Title: Prospective Evaluation of Image and Molecular Fingerprint Characterization to Guide Treatment With Tyrosine Kinase Inhibitors in Hepatocellular Carcinoma
Brief Title: Fingerprint Characterization Tyrosine Kinase Inhibitors in Advanced HCC
Acronym: e:Med-HCC-2
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment due to COVID-19 pandemic and several newly approved treatment options
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Michael Bitzer, Associate Director Internal Medicine I, University Hospital Tuebingen
Other Study IDs: e:Med-HCC-2
Record Dates: First submitted 2018-12-16; First posted 2019-05-22 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma; Sorafenib
Keywords: Liver Cancer; Imaging; Molecular Charakterization; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor Biopsy, Circulating DNA, PBMCs, Circulating Metabolites
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sorafenib treated HCC patients: No intervention is performed. This is an observational study.

SUMMARY:
This study is a prospective evaluation of a multiscale prediction model for the treatment with tyrosine kinase inhibitors (TKI) in HCC. Patients with HCC that qualify for systemic treatment with TKIs will be included. At baseline, prior to treatment, molecular and image fingerprints are collected (fingerprint #1). Further fingerprint investigations will be performed after a short treatment period at week 4 (fingerprint #2) and optional at tumor progression (Fingerprint #3). Based on previous findings from a preceding trial the fingerprint diagnostics #1 and #2 will be used to determine a prediction for treatment outcome at the earliest possible point in time ("therapy prediction"). This prediction will be compared to the prospectively determined outcome of the treated patients in this study (validation cohort; primary study endpoint). Fingerprint #3 will be optional to generate hypothesis for treatment failure.

DETAILED DESCRIPTION:
The aim of this prospective observational clinical study is to validate prognostic parameters for the treatment with tyrosine kinase inhibitors (TKI) that have been identified in a separate patient cohort with HCC (Study title "Fingerprint characterization of advanced HCC to optimize treatment decisions and enable an early prediction of therapy resistance", ClinicalTrials.gov Identifier NCT02372162). Based on these previous findings, predefined parameters that have been found to correlate with therapy responses will be determined for the patients in this observational trial. Diagnostic procedures include an image fingerprint (MRI and multi-phase CT scan of tumor manifestations, radiomics analysis of defined tumor areas, ultrasound elastography and a molecular fingerprint with exome and transcriptome sequencing from tumor tissue, single cell sequencing of PBMCs, MR spectroscopy for metabolomics analysis of blood and urine. These parameters at baseline will be used to predict therapy outcome, which will be prospectively compared to the clinical outcome under treatment with sorafenib. A second fingerprint will be collected at 4 weeks treatment and optional at tumor progression. New hypothesis generating parameters will be investigated in this patient cohort .

ELIGIBILITY:
Inclusion Criteria:

1. HCC patients with indication for the treatment with an approved tyrosine kinase inhibitor, irrespective of previous systemic therapies.
2. If prior systemic therapies had been applied, progression has to be documented prior to the start of treatment.
3. Male or female ≥ 18 years and written informed consent.
4. Histologically confirmed advanced stage hepatocellular carcinoma, BCLC class B or C.
5. Child-Pugh class A or B. Only patients with Child-Pugh index class B of not more than 7 will be included. Patients with untreatable ascites or hepatic encephalopathy > Grade 1 are excluded (see exclusion criteria).
6. ECOG performance status 0, 1 or 2.
7. Life expectancy of 12 weeks or more.
8. At least one measurable lesion without previous local therapy and that is suitable for accurate repeated measurements as per mRECIST guidelines.
9. Adequate hematological parameters, as demonstrated by:
10. Hemoglobin ≥ 9.0 g/dl (SI units: 5.6 mmol/l);
11. WBC ≥ 2.5 x 109/l;
12. Platelets ≥ 60 x 109/l;
13. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 times upper limit of normal range (ULNR);
14. Bilirubin ≤ 3 mg/dl;
15. Serum creatinine ≤ 1.5 mg/dl (SI units: 132 µmol/l);
16. Prothrombin Time (PT) International Normalized Ratio (INR) ≤ 1.5.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for study participation:

1. Renal failure requiring hemo- or peritoneal dialysis.
2. Patients with no adequate treatment for gastrointestinal bleeding and esophagus varices within 14 days prior to study entry.
3. Child-Pugh index class B in combination with more than slight ascites or hepatic encephalopathy > Grade I.
4. Altered mental status precluding understanding of the informed consent process.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will prospectively enrol all patients with HCC at our institution that qualify for a systemic treatment with sorafenib that fulfil the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
To prospectively evaluate image fingerprint analysis of HCC tumor tissue to predict therapy responses | 6 months after therapy initiation
  MRI and CT scan, including radiomics analysis
To prospectively evaluate molecular fingerprint analysis of HCC tumor tissue to predict therapy responses | 6 months after therapy initiation
  Multiscale analysis of exome, transcriptome and metabolic Tumor characteristics

SECONDARY OUTCOMES:
Time needed to determine parameter based prediction of therapy outcome for single parameters and for multiscale modelling | Diagnostic procedures at baseline and between week 3 and 6 after treatment initiation
  Days needed for prediction of therapy outcome by image, molecular and metabolic analysis
Progression Free Survival | Median PFS is expected between 3.5 and 5.5 months
  Months
Radiologically determined time to tumor progression (TTP) | Median TTP is expected between 3.5 and 5.5 months
  Months
Objective response rate (ORR) as measured by the sum of partial and complete responders. | Within 6 months after treatment initiation
  % of all treated patients
Duration of tumor stabilization (CR, PR, SD) | Through study completion, up to 18 months
  Days of duration of CR, PR or SD after diagnosis of best response
Overall Survival (OS) | Current data suggest approximately 12 months
  Months
To prospectively assess patient-reported outcome of HCC patients under treatment with sorafenib | Through study completion, up to 18 months
  EORTC QLQ-C30 questionnaire
Distribution of sorafenib adverse drug reactions | Through study completion during sorafenib treatment, up to 18 months
  CTCAE criteria
Feasibility of detection of circulating miRNA | Baseline and between week 3 and 6 after treatment initiation
  Change of miRNA detection in peripheral blood sample between baseline and after treatment initiation
Changes of Radiomics analysis under treatment with Sorafenib | Baseline and between week 3 and 6 after treatment initiation
  Collection of radiomics features of tumor tissue at baseline and after treatment initiation
Changes of ultrasound elastography under treatment with Sorafenib | Baseline and between week 3 and 6 after treatment initiation
  Determination of ultrasound elastography of tumor tissue at baseline and after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bitzer, MD, Principal Investigator — University Hospital, Eberhard Kars University Tübingen; Nisar P Malek, MD, Principal Investigator — University Hospital, Eberhard Kars University Tübingen
Locations (1):
- University Hospital Eberhard Karls University, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No